CLINICAL TRIAL: NCT05617222
Title: The Impact of Bed Rest and Aging on Muscle Mass and Muscle Function: Effects of Neuromuscular Electrical Stimulation
Brief Title: The Impact of Bed Rest, Aging and NMES on Skeletal Muscle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Suetta, Professor, Dr.Med, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-20038614
Record Dates: First submitted 2022-08-22; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Disuse Atrophy (Muscle) of Lower Extremities; Muscle Function; Neuromuscular Electrical Stimulation; Myofibrillar Protein Synthesis
MeSH Terms: conditions — Muscular Disorders, Atrophic | interventions — Bed Rest

STUDY DESIGN:
Intervention Model Description: Participants are subjected to 5 days bed rest. One leg will receive 3/daily neuromuscular electrical stimulation. The contralateral leg will serve as control-leg undergo disuse only.
Who Masked: Outcomes Assessor
Masking Description: The assessors will be without knowledge of which leg has received neuromuscular electrical stimulation and which leg was control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bed rest- Control (Active Comparator): One leg will be subjected to disuse by bed rest and will not receive further treatment during the bed rest period.
  Interventions: Other: Bed rest
- Bed rest + NMES (Experimental): One leg will be subjected to disuse by bed rest and will in addition receive neuromuscular electrical stimulation of the quadriceps muscle 3 times/day.
  Interventions: Other: Bed rest; Other: Neuromuscular electrical stimulation

INTERVENTIONS:
Other: Bed rest — 5 days of strict bed rest
Other: Neuromuscular electrical stimulation — Unilateral neuromuscular electrical stimulation (m. Quadriceps)
  Arms: Bed rest + NMES

SUMMARY:
Loss of muscle mass is common phenotypic trait of muscular disuse and ageing. The loss of muscle mass affects, among others, the ability to maintain homeostasis of glucose metabolism and the energy reservoir in catabolic conditions, while also affecting mechanical muscle function which can cause detrimental impairments in general functional status and hence quality of life.

However, a limited amount of research has attempted to elucidate molecular regulators of muscle mass loss following bed rest in older individuals and across genders. Consequently, the mechanistic drivers are unresolved and there are currently no effective therapeutic strategies to counteract muscle wasting and loss of function in individuals submitted to bed rest e.g. during hospitalization.

Purpose The purpose is to examine the effects of 5 days of bed rest on muscle mass, including myofibrillar protein synthesis and breakdown, and muscle function, and elucidate molecular regulators of muscle mass loss and metabolic pathways, while also investigating if potential negative effects can be counteracted by daily NeuroMuscular Electrical Stimulation (NMES) across different age and genders.

Methods The study is designed as a randomized controlled cross-over 5-day bed rest study including a group of healthy young (18-30 years) and healthy old (65-80 years) men and women.

Participants will receive daily electrical stimulation (NMES) of the thigh muscles (30 min x 3/day) on one leg (ES), while the other leg serves as a control (CON).

Participants will be tested at baseline (pre) and after (post) intervention for muscle strength, muscle power, balance, and muscle activation. Blood samples are collected at several time points and muscle biopsies are sampled pre- and post-intervention along with assessment of whole-body muscle mass and thigh muscle mass.

Scientific exposition The results from the study can potentially provide insight into the adaptive mechanisms associated with NMES training and muscular disuse on both cellular- and whole-body level. The understanding of the underlying mechanisms is crucial for the application of NMES in a therapeutic context and will furthermore help us understand the basic mechanism regulating the skeletal muscle mass during both training and muscular disuse.

Overall, the results can potentially help establishing treatments to counteract loss of muscle mass, muscle function and muscle health during periods of muscular disuse.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age between 18-30 or 65-80 years
* Injury free in the lower extremities (No previous or current knee injuries or knee pain)
* Normal weight
* Consumes normal diet

Exclusion Criteria:

* Cognitive impairment affecting the ability to participate in the study.
* Health related contraindications to participating in the intervention (i.e., bed rest and/or NMES), such as eczema and rash on the lower extremities
* Smoker
* Obesity
* Not able to speak or understand Danish.
* Acute or chronic diseases such as diabetes, cancer, embolism, infection, cardio-vascular diseases
* Use of medication which affects myofibrillar protein synthesis or the skeletal muscle tissue
* Use of other medication (e.g. anticoagulants, adrenal cortex hormone [within the last 3 months] etc.)
* Previous or current use of anabolic steroids
* Previous participation in research trials involving deuterium oxide or another stable isotope tracer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Myofiber cross-sectional area | Change from baseline after bed rest intervention
  Histochemical analysis of type I and type II myofiber cross-sectional area
Assessment of myofibrillar protein synthesis | Assessed during the period from pre-intervention biopsies (day 0, first day of bed rest) to post-intervention biopsies (day 5, last day and cessation of bed rest)
  Quantification of myofibrillar protein synthesis using the stable-isotope amino acid tracer deuterium oxide (D2O)
Change in maximal isometric muscle strength and superimposed twitch | Change from baseline after bed rest intervention
  Maximal isometric voluntary quadriceps strength combined with the superimposed twitch technique to assess maximal strength and voluntary muscle activation

SECONDARY OUTCOMES:
Change in total Akt protein assessed by Western blot | Change from baseline after bed rest intervention
  Assessment of Akt protein by Western Blot analysis using muscle tissue from vastus lateralis
Change in total mTOR protein assessed by Western blot | Change from baseline after bed rest intervention
  Assessment of mTOR protein by Western Blot analysis using muscle tissue from vastus lateralis
Change in total MuRF-1 protein assessed by Western blot | Change from baseline after bed rest intervention
  Assessment of MuRF-1 protein by Western Blot analysis using muscle tissue from vastus lateralis
Change in total Atrogin-1 protein assessed by Western blot | Change from baseline after bed rest intervention
  Assessment of Atrogin-1 protein by Western Blot analysis using muscle tissue from vastus lateralis
Change in total myostatin protein assessed by Western blot | Change from baseline after bed rest intervention
  Assessment of myostatin protein by Western Blot analysis using muscle tissue from vastus lateralis
Change in quadriceps muscle morphology and architecture by ultrasound scan | Change from baseline after bed rest intervention
  Ultrasound scan of rectus femoris and vastus lateralis muscle thickness and of vastus lateralis pennation angle
Change in body composition by DEXA scan | Change from baseline after bed rest intervention
  Assessment of whole body and regional lean mass and fat
Change in leg extensor power | Change from baseline after bed rest intervention
  Muscle power of the lower extremities assessed using the Nottingham power rig
Change in sway - postural balance | Change from baseline after bed rest intervention
  Measurement of displacement of center of pressure during unilateral and bilateral stance
Change in triglycerides | Day 0, day 2, day 4 and day 5
  Fasting blood samples are collected for analysis of triglycerides
Change in cholesterol | Day 0, day 2, day 4 and day 5
  Fasting blood samples are collected for later analysis of cholesterol
Change in C-reactive protein (CRP) | Day 0, day 2, day 4 and day 5
  Fasting blood samples are collected for analysis of CRP values

OTHER OUTCOMES:
Accelerometer data | 3 days prior to the intervention
  Collecting accelerometer data to quantify habitual activities prior to bed rest period
Accelerometer data | Throughout the 5 day intervention
  Collecting accelerometer data to monitor activity throughout the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Suetta, Professor, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark